CLINICAL TRIAL: NCT00914212
Title: A Functional Magnetic Resonance Imaging (fMRI) Study of the Reproducibility and the Effect of Sibutramine During Fasted and Fed Conditions in Healthy Overweight and Obese Men
Brief Title: A Functional Magnetic Resonance Imaging (fMRI) Study in Overweight and Obese Men (0000-103)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0000-103; 103; 2009_597
Record Dates: First submitted 2009-06-01; First posted 2009-06-04 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — sibutramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Sibutramine
  Interventions: Drug: Comparator: sibutramine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Single dose placebo to sibutramine in two of three treatment periods.
  Arms: 2
Drug: Comparator: sibutramine — Single dose sibutramine 30 mg (2 x 15 mg) in one of three treatment periods.
  Other Names: sibutramine
  Arms: 1

SUMMARY:
This study will determine whether BOLD-fMRI can be used to probe hunger and satiety states in healthy overweight or obese men and also whether fasted/fed fMRI signals can be modulated by sibutramine.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male between 18 and 45 years of age
* Subject has a body mass index (BMI) between 28 and 35 kg/m^2
* Subject does not weigh more than 140 kg (309 lbs) at the screening visit
* Subject is right-handed
* Subject is a non-smoker
* Subject is in generally good health
* Subject has normal or corrected to normal vision

Exclusion Criteria:

* Subject works a night shift within 3 days of each treatment visit
* Subject has permanent cosmetic or metallic objects in his body
* Subject has attention deficit hyperactivity disorder (ADHD)
* Subject has or had sleep apnea
* Subject has a history of neurological disorders
* Subject has a history of any clinically significant disease or condition
* Subject is vegan or vegetarian
* Subject has a history of eating disorders
* Subject has had previous bariatric surgery

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Average percent signal change of the top 20% of activated voxels (AvgPSC20) during the fasted condition over six primary brain regions of interest (ROI) | Day 1

SECONDARY OUTCOMES:
Intraclass coefficient of correlation of the AvgPSC20 assessed during the fed and fasted conditions over the six ROIs | Day 1
Regional cerebral blood flow (rCBF) during the fasted condition with placebo or sibutramine in the six ROIs | Day 1
AvgPSC20 in the fed condition with placebo or sibutramine in the six ROIs | Day 1
Difference in PSC20 during fasted and fed conditions with placebo or sibutramine in the six ROIs | Day 1
rCBF during the fed condition with placebo or sibutramine in the six ROIs | Day 1
Difference in rCBF during fasted and fed conditions with placebo or sibutramine in the six ROIs | Day 1
Test-retest reliability of rCBF in the six ROIs during the fasted and fed states in men receiving placebo | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC